CLINICAL TRIAL: NCT03235310
Title: ANRS CO1 EPF Prospective Observational Cohort Study on Mother-to-child Transmission HIV1 and/or HIV2 and Prevention
Brief Title: Prospective Observational Cohort Study on Mother to Child Transmission HIV1/HIV2 and Prevention
Acronym: EPF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Other Study IDs: ANRS-CO1-EPF
Record Dates: First submitted 2016-09-29; First posted 2017-08-01 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Mother to Child Transmission of HIV
Keywords: HIV; Pregnancy; Prevention of mother-to-child transmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3 mL whole blood 3mL plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe over time the rate of mother to child transmission of HIV and its prevention (PMTCT), to identify risk factors for transmission and to evaluate the safety of PMTCT strategies on outcome of pregnancy and in children not infected with HIV

DETAILED DESCRIPTION:
The CO1-EPF prospectively enrolled HIV-infected women who deliver in 25 centers throughout France, except in case of refusal.

Maternal clinical, biological and therapeutic data before and during pregnancy are collected at delivery. The children are examined clinically and biologically at birth, 1, 3, 6, 12 and 24 months. An infant is considered as non infected if two virologic tests are negative beyond the prophylactic treatment or serology is negative after 18 months. An infant is considered as infected if HIV1 is detected by virologic tests on two occasions (polymerase chain reactions, viral culture or p24 antigenemia) and if anti-HIV1 antibodies (ELISA and Western blot) persist after 18 months of age. Follow up is stopped at 24 months for uninfected infants whereas infected infants are enrolled in the CO10 EPF paediatric cohort. No specific recommendation for HIV treatment and obstetrical care are made for women and children included in the cohort, although national guidelines for prevention of MTCT are regularly published and updated. Frozen maternal samples blood and plasma are stored in a centralized laboratory. A research of patients patients lost to follow-up (last visit <24 months) and monitoring is performed regularly in all sites.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women >= 18 years
* infected with HIV1 and/or HIV2

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion as soon as possible during pregnancy of HIV-women in the largest obstetrical sites (17 in Paris area and 8 elsewhere in mainland France)
Sampling Method: Non-Probability Sample
Enrollment: 18200 (Estimated)
Dates: Start 1997-07; Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PMTCT strategies by measuring rate of mother to child transmission of HIV | At birth, 1 month, 3 months, 6 months, 12 months and 18-24 months
  Number of infected children (HIV RNA >50c/mL or Positive serology) reported on the total number of children

SECONDARY OUTCOMES:
Immuno-virological response during pregnancy | At inclusion up to childbirth
  HIV ARN <50c/mL, CD4 cells count>500 cells/mL
Tolerance and toxicity of different kind of MTCT prophylaxis during pregnancy | At inclusion up to childbirth
  incidence of pathologies during pregnancy (Number of cases of preeclampsia, Number of cases of cholestasis, CDC stage)
Impact of different kind of MTCT prophylaxis on childbirth | At delivery
  Childbirth mode (Number of emergency Caesarean section, Number of planned caesarean section)
Impact of different kind of MTCT prophylaxis during pregnancy on uninfected children | At childbirth, 1 month, 3 months, 6 months, 12 months and 18-24 months
  Clinical abnormalities (occurrence of adverse events)
Risk of mother-to-child transmission of VHC, VHB and CMV co-infections | At birth, 6 months, 12 months and 18-24 months
  Hepatitis B serology positive, Hepatitis C serology positive, presence of CMV in the urine

CONTACTS AND LOCATIONS:
Overall Officials: Josiane Warszawski, Principal Investigator — CESP INSERM U1018
Locations (28):
- France (28):
  - Centre Hospitalier Victor Dupuy, Argenteuil
  - Hôpital Jean Verdier, Bondy
  - Hôpital Antoine Béclère, Clamart
  - Hôpital de Beaujon, Clichy
  - Hôpital Louis Mourrier, Colombes
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Centre Hospitalier Intercommunal, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHR Jeanne de Flandres, Lille
  - Hôpital de La Croix Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Femme Mère Enfant, Lyon
  - Hôpital de la conception, Marseille
  - CHR Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Intercommunal, Montreuil
  - Hôtel Dieu, Nantes
  - CHU Hôpital de l'Archet II, Nice
  - Groupe Hospitalier Cochin Tarnier Port-Royal, Paris
  - Groupe Hospitalier Necker, Paris
  - Groupe Hospitalier Pitié Salpêtrière, Paris
  - Hôpital Bichat- Claude Bernard, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Tenon, Paris
  - Hôpital Trousseau, Paris
  - Centre Hospitalier Général- Hôpital Delafontaine, Saint-Denis
  - Hôpital Civil / Hôpital de Haute Pierre, Strasbourg
  - CHU Paule de Viguier, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mandelbrot L, Tubiana R, Le Chenadec J, Dollfus C, Faye A, Pannier E, Matheron S, Khuong MA, Garrait V, Reliquet V, Devidas A, Berrebi A, Allisy C, Elleau C, Arvieux C, Rouzioux C, Warszawski J, Blanche S; ANRS-EPF Study Group. No perinatal HIV-1 transmission from women with effective antiretroviral therapy starting before conception. Clin Infect Dis. 2015 Dec 1;61(11):1715-25. doi: 10.1093/cid/civ578. Epub 2015 Jul 21. PMID 26197844
- [Result] Taron-Brocard C, Le Chenadec J, Faye A, Dollfus C, Goetghebuer T, Gajdos V, Labaune JM, Perilhou A, Mandelbrot L, Blanche S, Warszawski J; France REcherche Nord&Sud Sida-HIV Hepatites - Enquete Perinatale Francaise - CO1/CO11 Study Group. Increased risk of serious bacterial infections due to maternal immunosuppression in HIV-exposed uninfected infants in a European country. Clin Infect Dis. 2014 Nov 1;59(9):1332-45. doi: 10.1093/cid/ciu586. Epub 2014 Jul 22. PMID 25053719
- [Result] Sibiude J, Mandelbrot L, Blanche S, Le Chenadec J, Boullag-Bonnet N, Faye A, Dollfus C, Tubiana R, Bonnet D, Lelong N, Khoshnood B, Warszawski J. Association between prenatal exposure to antiretroviral therapy and birth defects: an analysis of the French perinatal cohort study (ANRS CO1/CO11). PLoS Med. 2014 Apr 29;11(4):e1001635. doi: 10.1371/journal.pmed.1001635. eCollection 2014 Apr. PMID 24781315
- [Result] Briand N, Jasseron C, Sibiude J, Azria E, Pollet J, Hammou Y, Warszawski J, Mandelbrot L. Cesarean section for HIV-infected women in the combination antiretroviral therapies era, 2000-2010. Am J Obstet Gynecol. 2013 Oct;209(4):335.e1-335.e12. doi: 10.1016/j.ajog.2013.06.021. Epub 2013 Jun 18. PMID 23791563
- [Result] Briand N, Warszawski J, Mandelbrot L, Dollfus C, Pannier E, Cravello L, Nguyen R, Matheron I, Winer N, Tubiana R, Rouzioux C, Faye A, Blanche S; ANRS-EPF CO1-CO11 Study Group. Is intrapartum intravenous zidovudine for prevention of mother-to-child HIV-1 transmission still useful in the combination antiretroviral therapy era? Clin Infect Dis. 2013 Sep;57(6):903-14. doi: 10.1093/cid/cit374. Epub 2013 May 31. PMID 23728147
- [Result] Rachas A, Warszawski J, Le Chenadec J, Legeai C, Teglas JP, Goujard C, Rouzioux C, Mandelbrot L, Tubiana R, Meyer L. Does pregnancy affect the early response to cART? AIDS. 2013 Jan 28;27(3):357-67. doi: 10.1097/QAD.0b013e32835ac8bc. PMID 23079802
- [Result] Jasseron C, Mandelbrot L, Dollfus C, Trocme N, Tubiana R, Teglas JP, Faye A, Rouzioux C, Blanche S, Warszawski J. Non-disclosure of a pregnant woman's HIV status to her partner is associated with non-optimal prevention of mother-to-child transmission. AIDS Behav. 2013 Feb;17(2):488-97. doi: 10.1007/s10461-011-0084-y. PMID 22130651
- [Result] Simon A, Warszawski J, Kariyawasam D, Le Chenadec J, Benhammou V, Czernichow P, Foissac F, Laborde K, Treluyer JM, Firtion G, Layouni I, Munzer M, Bavoux F, Polak M, Blanche S; ANRS French Perinatal Cohort Study Group. Association of prenatal and postnatal exposure to lopinavir-ritonavir and adrenal dysfunction among uninfected infants of HIV-infected mothers. JAMA. 2011 Jul 6;306(1):70-8. doi: 10.1001/jama.2011.915. PMID 21730243
- [Result] Sibiude J, Warszawski J, Tubiana R, Dollfus C, Faye A, Rouzioux C, Teglas JP, Ekoukou D, Blanche S, Mandelbrot L. Premature delivery in HIV-infected women starting protease inhibitor therapy during pregnancy: role of the ritonavir boost? Clin Infect Dis. 2012 May;54(9):1348-60. doi: 10.1093/cid/cis198. Epub 2012 Mar 28. PMID 22460969
- [Result] Tubiana R, Le Chenadec J, Rouzioux C, Mandelbrot L, Hamrene K, Dollfus C, Faye A, Delaugerre C, Blanche S, Warszawski J. Factors associated with mother-to-child transmission of HIV-1 despite a maternal viral load <500 copies/ml at delivery: a case-control study nested in the French perinatal cohort (EPF-ANRS CO1). Clin Infect Dis. 2010 Feb 15;50(4):585-96. doi: 10.1086/650005. PMID 20070234
- [Result] Briand N, Mandelbrot L, Le Chenadec J, Tubiana R, Teglas JP, Faye A, Dollfus C, Rouzioux C, Blanche S, Warszawski J; ANRS French Perinatal Cohort. No relation between in-utero exposure to HAART and intrauterine growth retardation. AIDS. 2009 Jun 19;23(10):1235-43. doi: 10.1097/QAD.0b013e32832be0df. PMID 19424054
- [Result] Mandelbrot L, Jasseron C, Ekoukou D, Batallan A, Bongain A, Pannier E, Blanche S, Tubiana R, Rouzioux C, Warszawski J; ANRS French Perinatal Cohort (EPF). Amniocentesis and mother-to-child human immunodeficiency virus transmission in the Agence Nationale de Recherches sur le SIDA et les Hepatites Virales French Perinatal Cohort. Am J Obstet Gynecol. 2009 Feb;200(2):160.e1-9. doi: 10.1016/j.ajog.2008.08.049. Epub 2008 Nov 4. PMID 18986640
- [Result] Jasseron C, Mandelbrot L, Tubiana R, Teglas JP, Faye A, Dollfus C, Le Chenadec J, Rouzioux C, Blanche S, Warszawski J; ANRS French Perinatal Cohort. Prevention of mother-to-child HIV transmission: similar access for sub-Sahara African immigrants and for French women? AIDS. 2008 Jul 31;22(12):1503-11. doi: 10.1097/QAD.0b013e3283065b8c. PMID 18614874
- [Result] Benhammou V, Warszawski J, Bellec S, Doz F, Andre N, Lacour B, Levine M, Bavoux F, Tubiana R, Mandelbrot L, Clavel J, Blanche S; ANRS-Enquete Perinatale Francaise. Incidence of cancer in children perinatally exposed to nucleoside reverse transcriptase inhibitors. AIDS. 2008 Oct 18;22(16):2165-77. doi: 10.1097/QAD.0b013e328311d18b. PMID 18832880
- [Result] Warszawski J, Tubiana R, Le Chenadec J, Blanche S, Teglas JP, Dollfus C, Faye A, Burgard M, Rouzioux C, Mandelbrot L; ANRS French Perinatal Cohort. Mother-to-child HIV transmission despite antiretroviral therapy in the ANRS French Perinatal Cohort. AIDS. 2008 Jan 11;22(2):289-99. doi: 10.1097/QAD.0b013e3282f3d63c. PMID 18097232